CLINICAL TRIAL: NCT01035671
Title: A Phase 2a, Double-Blind, Randomized, Placebo-Controlled, 28 Day, Three-arm, Parallel Group Study of A0001 in the Treatment of Subjects With Friedreich's Ataxia
Brief Title: Safety and Efficacy Study of A0001 in Subjects With Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penwest Pharmaceuticals Co. (Industry)
Responsible Party: Thomas Sciascia, MD/Chief Medical Officer and VP Clinical Operations and Regulatory Affairs, Penwest Pharmaceuticals Co.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRD02
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — tocopherylquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental): A0001 (0.5 g BID)
  Interventions: Drug: alpha-tocopherolquinone (A0001)
- High Dose (Experimental): A0001 (0.75 g BID)
  Interventions: Drug: alpha-tocopherolquinone (A0001)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alpha-tocopherolquinone (A0001) — 28 days of low dose (1.0 g total daily dose) oral A0001 capsules. Treatment taken twice daily with meals.
  Arms: Low Dose
Drug: alpha-tocopherolquinone (A0001) — 28 days of high dose (1.5 g total daily dose) oral A0001 capsules. Treatment taken twice daily with meals.
  Arms: High Dose
Drug: placebo — 28 days of placebo oral capsules. Treatment taken twice daily with meals.
  Arms: Placebo

SUMMARY:
This is a Phase 2a double-blind, placebo-controlled study with two dose levels of A0001 given twice daily for 28 days. Potential subjects will be screened first to determine eligibility, after which they will be randomized to receive either a high dose of A0001, a low dose of A0001 or placebo for 28 days.

Eligible subjects will return within 21 days of screening for the baseline visit and randomization to one of three potential treatments. The subjects will be required to take 3 capsules of study medication in the morning with a morning meal and 3 capsules of study medication at night with an evening meal for 28 days. Additional visits to the clinic are planned for Day 14 and Day 28, at which time a number of clinical and biochemical assessments will be done.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with genetically confirmed Friedreich's Ataxia (GAA or point mutation)
* Impaired Glucose Tolerance, measured by Oral GTT

Exclusion Criteria:

* Overt Diabetes Mellitus
* Presence of clinically significant cardiovascular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in Disposition Index of Glucose Regulation, determined by Frequent Sampling IV Glucose Tolerance Test | Baseline, Day 14 and Day 28

SECONDARY OUTCOMES:
Sensitivity index (SI) calculated from IVGTT | Baseline, Day 14 and Day 28
Glucose effectiveness (SG) calculated from IVGTT | Baseline, Day 14 and Day 28
AIRg for glucose and insulin during IVGTT | Baseline, Day 14 and Day 28
Fasting Glucose, Insulin and Lactate | Baseline, Day 14 and Day 28
HbA1C | Baseline, Day 14 and Day 28
Plasma 1,5-anhydroglucitol (1,5-AG) (Glycomark) | Baseline, Day 14 and Day28
Specific Activity of Complex 1 in whole blood | Baseline, Day 14 and Day 28
Timed 25 Foot Walk Test | Baseline and Day 28
FARS/neurological exam | Baseline and Day 28
9-Hole Peg Test | Baseline, Day 14 and Day 28
Vision Low Contrast Letter Acuity Test | Baseline and Day 28
Global Impression of Clinical Severity | Baseline, Day 14 and Day 28
Modified Fatigue Impact Scale | Baseline and Day 28
Activities of Daily Living | Baseline and Day 28
SF-36® | Baseline and Day 28

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lynch DR, Willi SM, Wilson RB, Cotticelli MG, Brigatti KW, Deutsch EC, Kucheruk O, Shrader W, Rioux P, Miller G, Hawi A, Sciascia T. A0001 in Friedreich ataxia: biochemical characterization and effects in a clinical trial. Mov Disord. 2012 Jul;27(8):1026-33. doi: 10.1002/mds.25058. Epub 2012 Jun 28. PMID 22744651
- [Derived] Friedman LS, Schadt KA, Regner SR, Mark GE, Lin KY, Sciascia T, St John Sutton M, Willi S, Lynch DR. Elevation of serum cardiac troponin I in a cross-sectional cohort of asymptomatic subjects with Friedreich ataxia. Int J Cardiol. 2013 Aug 20;167(4):1622-4. doi: 10.1016/j.ijcard.2012.04.159. Epub 2012 May 26. PMID 22633670